CLINICAL TRIAL: NCT02939339
Title: Theta Burst TMS as a Tool to Change Smoking Behavior
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00042165
Record Dates: First submitted 2016-09-01; First posted 2016-10-20 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Smoking; Addiction
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Smoking; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- real treatment (Experimental): continuous theta burst stimulation (real) will be delivered
  Interventions: Device: continuous theta burst stimulation (real)
- sham treatment (Sham Comparator): continuous theta burst stimulation (sham) will be delivered
  Interventions: Device: continuous theta burst stimulation (sham)

INTERVENTIONS:
Device: continuous theta burst stimulation (real) — a form of transcranial magnetic stimulation that noninvasively induces a depression in brain reactivity
  Other Names: cTBS (active)
  Arms: real treatment
Device: continuous theta burst stimulation (sham) — a sham version of a form of transcranial magnetic stimulation that noninvasively induces a depression in brain reactivity
  Other Names: cTBS (sham)
  Arms: sham treatment

SUMMARY:
The goal of this study is to determine whether transcranial magnetic stimulation (TMS) is an effective treatment in decreasing craving in individuals who habitually smoke cigarettes. The study consists of six total visits to MUSC; one for the consent process, two that will include MRI scans, and five that will include TMS administration. Compensation will be provided for each visit.

DETAILED DESCRIPTION:
Prior and recent evidence suggests a role of medial prefrontal cortex (mPFC) in cigarette smoking. The present study will examine whether a five-day regimen of theta-burst transcranial magnetic stimulation (TMS) reduces cigarette smoking outside of the lab (examined through self-report and physiological measures) and motivation to smoke inside the lab (examined through behavioral tasks and functional MRI).

ELIGIBILITY:
Inclusion Criteria:

* smoke at least 10 cigarettes a day (on average)

Exclusion Criteria:

* comorbid mental or physical illness (managed or unmanaged)
* pregnancy
* use of prescription medication that might affect smoking or nicotine metabolism,
* use of smokeless tobacco or alternative nicotine products
* use illicit drugs of abuse (verified through urine screen and self-report),
* score of above a 7 on the Alcohol Use Disorders Identification Test (indicative of non-risky use),
* a history of epilepsy or seizures not otherwise specified (other than childhood febrile seizures)
* a history of chronic migraines,
* failure to meet all criteria on a standardized MRI/TMS safety screen (including but not limited to implanted electronic devices, bullets or metallic fragments above the waist, hair clips and piercings above the waist that cannot be removed)
* presence of any barriers to making contact between the TMS coil and the skin (e.g. cornrows that cannot be removed, glasses that the participant is unwilling to remove).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Percent BOLD signal change in the MPFC | immediately after the treatment
  The effect of real vs. sham cTBS to the leftt MPFC as a tool to modulate the brain response to craving will be assessed by comparing the brain activity in the limbic circuit before and after TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Hanlon, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinha R. New findings on biological factors predicting addiction relapse vulnerability. Curr Psychiatry Rep. 2011 Oct;13(5):398-405. doi: 10.1007/s11920-011-0224-0. PMID 21792580
- [Background] Kalivas PW, Volkow ND. The neural basis of addiction: a pathology of motivation and choice. Am J Psychiatry. 2005 Aug;162(8):1403-13. doi: 10.1176/appi.ajp.162.8.1403. PMID 16055761
- [Background] Sinha R, Catapano D, O'Malley S. Stress-induced craving and stress response in cocaine dependent individuals. Psychopharmacology (Berl). 1999 Mar;142(4):343-51. doi: 10.1007/s002130050898. PMID 10229058
- [Background] Lee JL, Milton AL, Everitt BJ. Cue-induced cocaine seeking and relapse are reduced by disruption of drug memory reconsolidation. J Neurosci. 2006 May 31;26(22):5881-7. doi: 10.1523/JNEUROSCI.0323-06.2006. PMID 16738229
- [Background] Volkow ND, Wang GJ, Fowler JS, Tomasi D. Addiction circuitry in the human brain. Annu Rev Pharmacol Toxicol. 2012;52:321-36. doi: 10.1146/annurev-pharmtox-010611-134625. Epub 2011 Sep 27. PMID 21961707
- [Background] Bolla K, Ernst M, Kiehl K, Mouratidis M, Eldreth D, Contoreggi C, Matochik J, Kurian V, Cadet J, Kimes A, Funderburk F, London E. Prefrontal cortical dysfunction in abstinent cocaine abusers. J Neuropsychiatry Clin Neurosci. 2004 Fall;16(4):456-64. doi: 10.1176/jnp.16.4.456. PMID 15616172
- [Background] Bolla KI, Eldreth DA, London ED, Kiehl KA, Mouratidis M, Contoreggi C, Matochik JA, Kurian V, Cadet JL, Kimes AS, Funderburk FR, Ernst M. Orbitofrontal cortex dysfunction in abstinent cocaine abusers performing a decision-making task. Neuroimage. 2003 Jul;19(3):1085-94. doi: 10.1016/s1053-8119(03)00113-7. PMID 12880834
- [Background] Hanlon CA, Wesley MJ, Stapleton JR, Laurienti PJ, Porrino LJ. The association between frontal-striatal connectivity and sensorimotor control in cocaine users. Drug Alcohol Depend. 2011 Jun 1;115(3):240-3. doi: 10.1016/j.drugalcdep.2010.11.008. Epub 2010 Dec 28. PMID 21193273
- [Background] Gu H, Salmeron BJ, Ross TJ, Geng X, Zhan W, Stein EA, Yang Y. Mesocorticolimbic circuits are impaired in chronic cocaine users as demonstrated by resting-state functional connectivity. Neuroimage. 2010 Nov 1;53(2):593-601. doi: 10.1016/j.neuroimage.2010.06.066. Epub 2010 Jul 11. PMID 20603217
- [Background] Bear MF, Malenka RC. Synaptic plasticity: LTP and LTD. Curr Opin Neurobiol. 1994 Jun;4(3):389-99. doi: 10.1016/0959-4388(94)90101-5. PMID 7919934
- [Background] Malenka RC, Bear MF. LTP and LTD: an embarrassment of riches. Neuron. 2004 Sep 30;44(1):5-21. doi: 10.1016/j.neuron.2004.09.012. PMID 15450156
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Di Lazzaro V, Pilato F, Saturno E, Oliviero A, Dileone M, Mazzone P, Insola A, Tonali PA, Ranieri F, Huang YZ, Rothwell JC. Theta-burst repetitive transcranial magnetic stimulation suppresses specific excitatory circuits in the human motor cortex. J Physiol. 2005 Jun 15;565(Pt 3):945-50. doi: 10.1113/jphysiol.2005.087288. Epub 2005 Apr 21. PMID 15845575
- [Background] Verbruggen F, Aron AR, Stevens MA, Chambers CD. Theta burst stimulation dissociates attention and action updating in human inferior frontal cortex. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13966-71. doi: 10.1073/pnas.1001957107. Epub 2010 Jul 14. PMID 20631303
- [Background] Cho SS, Ko JH, Pellecchia G, Van Eimeren T, Cilia R, Strafella AP. Continuous theta burst stimulation of right dorsolateral prefrontal cortex induces changes in impulsivity level. Brain Stimul. 2010 Jul;3(3):170-6. doi: 10.1016/j.brs.2009.10.002. Epub 2009 Oct 31. PMID 20633446
- [Background] Jacobson L, Javitt DC, Lavidor M. Activation of inhibition: diminishing impulsive behavior by direct current stimulation over the inferior frontal gyrus. J Cogn Neurosci. 2011 Nov;23(11):3380-7. doi: 10.1162/jocn_a_00020. Epub 2011 Mar 31. PMID 21452949
- [Background] Camprodon JA, Martinez-Raga J, Alonso-Alonso M, Shih MC, Pascual-Leone A. One session of high frequency repetitive transcranial magnetic stimulation (rTMS) to the right prefrontal cortex transiently reduces cocaine craving. Drug Alcohol Depend. 2007 Jan 5;86(1):91-4. doi: 10.1016/j.drugalcdep.2006.06.002. Epub 2006 Sep 12. PMID 16971058
- [Background] Politi E, Fauci E, Santoro A, Smeraldi E. Daily sessions of transcranial magnetic stimulation to the left prefrontal cortex gradually reduce cocaine craving. Am J Addict. 2008 Jul-Aug;17(4):345-6. doi: 10.1080/10550490802139283. No abstract available. PMID 18612892
- [Background] Barr MS, Fitzgerald PB, Farzan F, George TP, Daskalakis ZJ. Transcranial magnetic stimulation to understand the pathophysiology and treatment of substance use disorders. Curr Drug Abuse Rev. 2008 Nov;1(3):328-39. doi: 10.2174/1874473710801030328. PMID 19630729
- [Background] Wing VC, Barr MS, Wass CE, Lipsman N, Lozano AM, Daskalakis ZJ, George TP. Brain stimulation methods to treat tobacco addiction. Brain Stimul. 2013 May;6(3):221-30. doi: 10.1016/j.brs.2012.06.008. Epub 2012 Jul 9. PMID 22809824
- [Background] Hanlon CA, Canterberry M, Taylor JJ, DeVries W, Li X, Brown TR, George MS. Probing the frontostriatal loops involved in executive and limbic processing via interleaved TMS and functional MRI at two prefrontal locations: a pilot study. PLoS One. 2013 Jul 9;8(7):e67917. doi: 10.1371/journal.pone.0067917. Print 2013. PMID 23874466
- [Background] Bestmann S, Baudewig J, Siebner HR, Rothwell JC, Frahm J. Functional MRI of the immediate impact of transcranial magnetic stimulation on cortical and subcortical motor circuits. Eur J Neurosci. 2004 Apr;19(7):1950-62. doi: 10.1111/j.1460-9568.2004.03277.x. PMID 15078569
- [Background] Bohning DE, Shastri A, Lomarev MP, Lorberbaum JP, Nahas Z, George MS. BOLD-fMRI response vs. transcranial magnetic stimulation (TMS) pulse-train length: testing for linearity. J Magn Reson Imaging. 2003 Mar;17(3):279-90. doi: 10.1002/jmri.10271. PMID 12594717
- [Background] Fox MD, Buckner RL, White MP, Greicius MD, Pascual-Leone A. Efficacy of transcranial magnetic stimulation targets for depression is related to intrinsic functional connectivity with the subgenual cingulate. Biol Psychiatry. 2012 Oct 1;72(7):595-603. doi: 10.1016/j.biopsych.2012.04.028. Epub 2012 Jun 1. PMID 22658708
- [Background] Vernet M, Bashir S, Yoo WK, Oberman L, Mizrahi I, Ifert-Miller F, Beck CJ, Pascual-Leone A. Reproducibility of the effects of theta burst stimulation on motor cortical plasticity in healthy participants. Clin Neurophysiol. 2014 Feb;125(2):320-6. doi: 10.1016/j.clinph.2013.07.004. Epub 2013 Aug 7. PMID 23932365
- [Background] Wilcox CE, Teshiba TM, Merideth F, Ling J, Mayer AR. Enhanced cue reactivity and fronto-striatal functional connectivity in cocaine use disorders. Drug Alcohol Depend. 2011 May 1;115(1-2):137-44. doi: 10.1016/j.drugalcdep.2011.01.009. Epub 2011 Apr 3. PMID 21466926
- [Background] Prisciandaro JJ, McRae-Clark AL, Myrick H, Henderson S, Brady KT. Brain activation to cocaine cues and motivation/treatment status. Addict Biol. 2014 Mar;19(2):240-9. doi: 10.1111/j.1369-1600.2012.00446.x. Epub 2012 Mar 28. PMID 22458561
- [Background] Borckardt JJ, Nahas Z, Koola J, George MS. Estimating resting motor thresholds in transcranial magnetic stimulation research and practice: a computer simulation evaluation of best methods. J ECT. 2006 Sep;22(3):169-75. doi: 10.1097/01.yct.0000235923.52741.72. PMID 16957531